CLINICAL TRIAL: NCT01098292
Title: Multidisciplinary Approach to the Study of Chronic Pelvic Pain: Trans-MAPP Control Study
Brief Title: Observational Study of Control Participants for the MAPP Research Network
Acronym: MAPP-Control
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 810668
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2013-05

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic
Keywords: Fibromyalgia; Irritable Bowel Syndrome; Chronic Fatigue Syndrome; Interstitial Cystitis; Chronic Prostatitis; Urological Chronic Pelvic Pain; Painful Bladder Syndrome
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Blood Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Control: Healthy Control participants do not suffer from any Urological Chronic Pelvic Pain Syndromes or from the following conditions:
  Fibromyalgia, Irritable Bowel Syndrome, Chronic Fatigue Syndrome
- Positive Control: Positive Control participants do not suffer from any Urological Pelvic Pain Syndromes like Interstitial Cystitis and/or Chronic Prostatitis. However Positive Controls have a history of one of the following conditions:
  Fibromyalgia, Irritable Bowel Syndrome, Chronic Fatigue Syndrome

SUMMARY:
The Control Study for the Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) Research Network has been established to focus on a broader approach to the study of Interstitial Cystitis (IC)/Painful Bladder Syndrome (PBS) in men and women, and Chronic Prostatitis (CP)/Chronic Pelvic Pain Syndrome (CPPS) in men, than previously undertaken.

Participants with no Urologic Pelvic Pain Syndromes as well as participants with specific conditions (Fibromyalgia (FM), Irritable Bowel Syndrome (IBS), Chronic Fatigue Syndrome (CFS)) are being recruited for the Trans-MAPP Control Study. These participants will act as a reference/control group for the Trans-MAPP Epidemiology & Phenotyping (EP) Study.

As with many chronic pain disorders, IC and CP are poorly understood, and treatment is often not helpful. The goal of this study is to better understand how pain is felt in people with IC or CP. The MAPP Control Study is an observational study that will enroll participants from 6 Discovery Sites and 3 Satellite Sites across the U.S. The investigators will ask questions and gather information about the health and life of the participants for research purposes. The investigators hope that this study will lead to improvement in the treatment of IC and CP.

DETAILED DESCRIPTION:
Trans-MAPP Control participants will only need to complete one study visit to collect baseline data and biospecimens. Potential participants will be scheduled for an eligibility screening session. Following screening, potentially eligible participants will complete a baseline phenotyping session, and biospecimen collections, which together are expected to take approximately 2.5 hours to complete. Participants will be provided with breaks as needed during the clinic visit.

ELIGIBILITY:
The eligibility criteria for both healthy controls and positive controls are based on the same set of criteria for the Urologic Chronic Pelvic Pain Syndrome (UCPPS) participants in the Trans-MAPP EP Study, with exception of additional criteria to exclude chronic pelvic pain symptoms and criteria to identify the co-morbid syndromes for the positive controls. All entry criteria are shown below; those specific to either healthy or positive control participants are so indicated.

Inclusion Criteria:

Participants are eligible for the Trans-MAPP Control Protocol if they meet the following general and gender-specific criteria listed below:

1. Participant has signed and dated the appropriate Informed Consent document.
2. Agreed to participate in Trans-MAPP Control Study procedures;

Inclusion Criteria for Healthy Controls only

1. Participant reports a response of "0" (zero) on the pain, pressure or discomfort scale.
2. Participant reports no chronic pain in the pelvic or bladder region, and reports chronic pain in no more than one other body region.
3. Participant reports no urological symptoms that have been evaluated, but are still present.

Inclusion Criteria for Positive Controls only:

1. Participant meets the validated criteria for one or more of the following conditions

1. Fibromyalgia (FM)
2. Irritable bowel syndrome (IBS)
3. Chronic fatigue syndrome (CFS)

Exclusion Criteria:

Individuals will not be eligible for enrollment in the Trans-MAPP Control Study if they meet any of the criteria:

1. Participant has an on-going symptomatic urethral stricture.
2. Participant has an on-going neurological disease or disorder affecting the bladder or bowel fistula.
3. Participant has a history of cystitis caused by tuberculosis or radiation therapy or Cytoxan/cyclophosphamide therapy.
4. Participant has augmentation cystoplasty or cystectomy.
5. Participant has a systemic autoimmune disorder (such as Crohn's Disease, Ulcerative Colitis, Lupus, Rheumatoid Arthritis, or Multiple Sclerosis).
6. Participant has a history of cancer (with the exception of skin cancer).
7. Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc).
8. Participant has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.

Exclusion Criteria for Males Only

1. Male participant diagnosed with unilateral orchialgia, without pelvic symptoms.
2. Male participant has a history of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, or prostate cryosurgery or laser procedure.

Exclusion Criteria for Females Only:

1) Female participant has a history of High-Grade Squamous Intraepithelial Lesion (HGSIL) / high-grade cervical dysplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Trans-MAPP Control Study population will include adult participants, at least 18 years of age, with no urological chronic pelvic pain syndromes. These participants will fall into two categories: Healthy Controls and Positive Controls.
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Baseline outcome measures | Baseline
  Extensive data on risk factors and outcomes measures will be collected for the Trans-MAPP Control Study. These measures can be classified into a number of primary domains as described below.
  1. General Measures of Sociodemographics, Health, and Quality of Life
  2. UCPPS Symptoms Measures
  3. Non-urological Symptom Measures
  4. Trait-like Personal Factors
  5. Biological Specimens

CONTACTS AND LOCATIONS:
Overall Officials: J. Quentin Clemens, MD, Study Chair — University of Michigan; Christopher Mullens, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: MAPP Research Network Website — http://mappnetwork.org